CLINICAL TRIAL: NCT07231224
Title: Postoperative Myofunctional Therapy Enhances Surgical Outcomes in Patients With Obstructive Sleep Apnea: A Prospective Comparative Stud
Brief Title: A Study of Myofunctional Therapy After Sleep Apnea Surgery
Acronym: MFT-OSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Collaborators: Taipei Medical University (Other); National Yang Ming Chiao Tung University Hospital (Other); National Tsing Hua University,Taiwan (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TMUJIRB No.201912067; W114YSR-03 (Other: Taipei Medical University Shuang Ho Hospital Young Scholar Research Grant); TMU113-AE1-B04 (Other: Taipei Medical University Newly Recruited Faculty Research Grant)
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Obstructive Sleep Apnea
Keywords: Obstructive sleep apnea; Myofunctional therapy (MFT); Upper airway surgery; Oropharyngeal exercises; Postoperative outcomes; Polysomnography (PSG); Apnea-Hypopnea Index (AHI)
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Myofunctional Therapy

STUDY DESIGN:
Intervention Model Description: Enrolled patients were divided into two parallel groups based on personal willingness after discussion: Group A (OP+MFT) or Group B (OP-only)
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OP+MFT Group (Experimental): Participants in this group underwent surgery and began a structured 12-week postoperative myofunctional therapy (MFT) program starting at the third postoperative week.
  Interventions: Procedure: myofunctional therapy
- OP-only Group (No Intervention): Participants in this group underwent the same surgical procedure but received only routine postoperative follow-up without any additional MFT training.

INTERVENTIONS:
Procedure: myofunctional therapy — A 12-week structured program of oropharyngeal exercises that commenced three weeks after surgery. The program consisted of initial face-to-face instruction, twice-daily home practice (15 minutes each) guided by videos, and biweekly supervision. Exercises included tongue elevation and protrusion drills, soft palate elevation, and pharyngeal wall contractions to enhance neuromuscular control of the upper airway.
  Arms: OP+MFT Group

SUMMARY:
Obstructive sleep apnea (OSA) is a common disorder characterized by recurrent upper airway collapse. While surgery is a common treatment, its success rates are variable. Myofunctional therapy (MFT), a program of targeted oropharyngeal exercises, has emerged as a promising adjunctive treatment to improve surgical outcomes.

This study prospectively compared outcomes in adult patients with moderate-to-severe OSA who received postoperative MFT (OP+MFT) versus those who underwent surgery alone (OP). Following surgery, patients were allocated to either the OP+MFT group, which began a 12-week MFT program, or the OP-only group. Polysomnography (PSG) was performed at baseline and at 3 and 12 months post-surgery.

The study found that the OP+MFT group showed significantly greater improvements in key sleep parameters, including the Apnea-Hypopnea Index (AHI) and lowest oxygen saturation, compared to the OP group. These benefits were most pronounced at the 3-month follow-up, supporting the conclusion that postoperative MFT is a safe and effective adjunct to surgery for OSA.

DETAILED DESCRIPTION:
Obstructive Sleep Apnea (OSA) is a prevalent condition associated with significant morbidity, including hypertension and cardiovascular disease. The first-line treatment, Continuous Positive Airway Pressure (CPAP), is limited by poor long-term patient adherence, with compliance rates often below 20%. For patients who are intolerant to CPAP, surgical options are available, but their long-term success rates are modest, averaging around 30%.

This study is based on the rationale that surgery primarily addresses static anatomical obstructions, while a key functional deficit-poor neuromuscular tone of the upper airway dilator muscles-remains uncorrected by surgery alone. Myofunctional therapy (MFT) is a structured exercise program designed to strengthen oropharyngeal muscles (e.g., tongue, soft palate), improve neuromuscular control, and enhance airway stability during sleep.

This study was designed to evaluate the synergistic effect of combining surgery with postoperative MFT. The hypothesis is that a dual approach, where surgery provides anatomical relief and MFT enhances dynamic airway stability, will lead to superior treatment outcomes compared to surgery alone.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-65 years
* Moderate-to-severe Obstructive Sleep Apnea (AHI ≥ 15 events/hour) confirmed by PSG
* Friedman palate position grade I-II and tonsil size grade III-IV
* Patients who refuse or are unable to tolerate CPAP

Exclusion Criteria:

* - Central or mixed sleep apnea
* BMI > 27 kg/m²
* Severe cardiopulmonary disease or psychiatric illness
* Pregnancy or cancer
* Significant weight gain during the follow-up period

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Change in Apnea-Hypopnea Index | Baseline, 3 months post-surgery, and 12 months post-surgery
  Change in AHI from baseline, measured by polysomnography in events per hour. Treatment success is defined as a reduction of ≥50% from baseline AHI and a final AHI of <20 events/hour.

SECONDARY OUTCOMES:
Change in Lowest Oxygen Saturation (LSaO₂) | Baseline, 3 months post-surgery, and 12 months post-surgery
  Change in the lowest oxygen saturation (LSaO₂) during sleep, measured by polysomnography as a percentage
Change in Snore Index | Baseline, 3 months post-surgery, and 12 months post-surgery
  Change in the snore index, measured by polysomnography as the percentage of total sleep time with snoring events

CONTACTS AND LOCATIONS:
Overall Officials: CHENGJUNG WU, MD, Principal Investigator — Shuang Ho Hospital, Taipei Medical University
Locations (1):
- Taipei Medical University - Shuang Ho Hospital, New Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
The data presented in this study are available on reasonable request from the corresponding author
Supporting Information: Study Protocol
Time Frame: Data will be available following the publication of the primary manuscript
Access Criteria: Data access can be granted upon reasonable request to the corresponding author. Requesters may need to provide a study protocol or analysis plan to ensure the responsible use of the de-identified data.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-01-07): https://cdn.clinicaltrials.gov/large-docs/24/NCT07231224/Prot_SAP_000.pdf
  • Informed Consent Form (2020-01-07): https://cdn.clinicaltrials.gov/large-docs/24/NCT07231224/ICF_001.pdf